CLINICAL TRIAL: NCT06460051
Title: Effects of Ultrasound-guided Maxillary Nerve Block Performed After Bimaxillary Osteotomy in Adult Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Servei Central d'Anestesiologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5TDGM
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Maxillary Diseases; Pain, Postoperative; Adult Patients Undergoing Bimaxillary Osteotomy
Keywords: Orthognatic surgery; Bimaxillary osteotomy; Maxillary nerve block; Ultrasound; Postoperative pain
MeSH Terms: conditions — Maxillary Diseases; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The researchers propose a double-blind (patient and nurse) prospective comparative experimental study. The patients included in the study will be scheduled for bimaxillary osteotomy and will be assigned consecutively and prospectively to one of the two groups (maxillary nerve block before surgery or block after surgery) with a plan to register up to 50 patients.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A 1:1 randomization table for patient allocation will be generated by a statistician who will not otherwise be involved in the study. Immediately upon the patient's arrival to the operating room, the research anesthesiologist will open a sealed, sequentially numbered opaque envelope containing the patient's assignment (block before surgery or block after surgery). Only anesthesiologists and operating room surgeons will not be blinded to patient assignment. This will be a double-blind study (patient and nurse). Patients will be unaware of the group they have been consecutively assigned to; and both the postoperative resuscitation nurses and the hospitalization ward nurses who will record visual analogue scale, analgesic consumption, onset of oral tolerance, postoperative nausea-vomiting and postoperative complications, will also be unaware of the analgesic treatment that the patient has received in the operating room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary nerve block before bimaxillary osteotomy (Active Comparator): Patients receive ultrasound-guided suprazigomatic maxillary nerve block after nasotracheal intubation before bimaxillary osteotomy.
  Interventions: Procedure: Maxillary nerve block
- Maxillary nerve block after bimaxillary osteotomy (Experimental): Patients receive ultrasound-guidedsuprazygomatic maxillary nerve block after bimaxillary osteotomy before extubation.
  Interventions: Procedure: Maxillary nerve block

INTERVENTIONS:
Procedure: Maxillary nerve block — Ultrasound-guided, suprazygomatic approach, infrazygomatic window
  Other Names: Ultrasound-guided maxillary nerve block

SUMMARY:
Bimaxillary osteotomy is a surgery procedure of the orthognathic surgery field for correction of dental and facial abnormalities, for both functional and aesthetic cases. The incidence of this abnormality is 5-10% of the population, and the etiology is unknown, with genetic, environmental and embryonic factors related. The surgery technic is complex, and requires osteotomy of the maxilla and jaw, which allows toward, forward, impact and rotation of these bones to fix the edges of the face. The anesthetic management of these patients is a challenge because of the difficult airway management and the perioperative pain control. Multimodal approach for pain control is a fact, and the use of local and regional anaesthesia is mandatory. The investigators propose bilateral ultrasound-guided suprazigomatic maxillary nerve block after bimaxillary osteotomy for a proper control of postoperative pain.

DETAILED DESCRIPTION:
Bimaxillary osteotomy is a surgical procedure in the field of orthognathic surgery (from Latin; "orthos" rectum and "gnathos" mandible) for the correction of dentofacial deformities, both for functional and aesthetic reasons. The incidence of this deformity is estimated to be in the order of 5-10% of the population; and its origin is still unknown, and genetic, environmental and embryonic factors are postulated. The surgical technique is complex, with the performance of mandibular and upper jaw osteotomies that allow these bones to be advanced, retracted, impacted and rotated, to align the facial axes. For all these reasons, the anesthetic management of these patients is a challenge. First, the foreseeable difficulty of managing the patient's airway; and second, the control of the patient's pain in the perioperative period.

Therefore, it is said that bimaxillary osteotomy is a frequent and potentially painful surgery in adults. Bimaxillary surgery under general anesthesia is common practice. And isolated non-ultrasound-guided peripheral nerve blocks and surgical field infiltration are widely used practices by surgeons. These minor blockages and infiltrations are used to avoid the unwanted effects of anesthetics and analgesics; particularly the adverse respiratory effects of opioids. The practice of loco-regional anesthesia therefore provides perioperative pain control in a multimodal way, showing effective postoperative analgesia and minimizing respiratory depression due to excessive use of opioids.

The introduction of loco-regional nerve blocks in the last three decades has meant a revolution in the management and control of perioperative pain for the anesthesiologist. The expansion of the practice of loco-regional nerve blocks has been seen in both the upper and lower limbs, as well as the trunk and abdomen. Conversely, facial blocks, superficial and deep, have not experienced the same; relegating its practice to the surgeon, or to the anesthesiologist who works in the field of chronic pain. The subsequent introduction of ultrasonography (USG) in the 1990s in the perioperative period was also an important advance for the anesthesiologist, both in terms of safety and in terms of ease of handling catheterizations of the venous and arterial lines, and the practice of loco-regional blocks.

Consequently, anesthesiologists already experienced at the USG have recently published on the use of ultrasound (US) for facial nerve block in children and adults undergoing maxillofacial surgery. USG devices are becoming more accessible, more portable, cheaper, and more secure; And therefore, its introduction in the field of perioperative pain management of maxillofacial surgery still has a long way to go.

The maxillary nerve, like the ophthalmic nerve, is only sensory. It is detached from the anterolateral border of the trigeminal ganglion, laterally to the ophthalmic. From its origin, it heads anteriorly, traverses the foramen round, and penetrates the background of the infratemporal fossa until it enters the pterygopalatine fossa (except for the middle meningeal nerve, all its branches reach the pterygopalatine fossa before reaching the facies). In the pterygopalatine fossa, the maxillary nerve is located at the top of the cavity and passes superiorly to the maxillary artery and superolaterally to the pterygopalatine ganglion. The maxillary nerve receives and conducts through its endings the sensitivity of the skin of the cheek, lower eyelid, wing of the nose and upper lip. Its deep branches conduct the sensitivity of the mucosa of the lower part of the nasal cavities or respiratory area, of the tooth roots and of the gums of the maxilla.

Therefore, in order to produce an effective anesthesia of the maxillary area, the anesthesiologists can introduce the needle through the pterygomaxillary fissure to the pterygopalatine fossa, with the risk of vascular and nerve puncture. But with the real-time view of ultrasound-guided block, these risks will be limited, allowing direct localization of the maxillary artery, needle position, and distribution of the LA within the pterygopalatine fossa. The pterygopalatine fossa is anatomically deep and surrounded by bones. The most optimal ultrasound window is the infrazygomatic pathway, allowing visualization of the entire axis of the pterygopalatine fossa up to the foramen round.

To carry out the maxillary nerve block, several approaches have been described. However, placing the ultrasound probe in an infrazygomatic position, and introducing the needle suprazygomaticly from the frontozygomatic angle is one of the safest and most recommended routes to reach the round foramen. This trajectory limits the insertion of the needle into the anterior portion of the foramen round, thus preventing inadvertent puncture of the intraorbital contents through the infraorbital fissure.

In general, in bimaxillary surgery it is the surgeon who performs the infiltrations with local anesthetic (AL) in a pre-incisional way to block the terminal branches of the maxillary nerve intraorally and intranasally. The choice of LA is influenced by considerations such as onset of action, duration, and toxicity. A wide range of LA have been used in maxillofacial surgery, such as lidocaine and bupivacaine, among others. The two LAs produce a reversible blockade of the sodium channel of the neuronal membrane, and are synthetic derivatives of cocaine. Both have three essential functional units (hydrophilic tertiary amide chain, linked by an intermediate amide chain to another lipophilic aromatic ring-portion). That is, they are both AL of the amide type; but even though they belong to the same group of LA, there are great differences in terms of initiation of action, duration of action and toxicity. Lidocaine has a faster onset of action (short latency) than bupivacaine, and has an antiarrhythmic effect. Bupivacaine is more potent and has a longer duration of action than lidocaine, although more cardiotoxic than other AL teams such as ropivacaine.

To date, the gold standard anesthetic technique has not been described, nor is the ideal time to perform it in patients who have undergone bimaxillary osteotomy surgery. The investigators now propose the performance of bilateral maxillary nerve block ultrasounded by suprazygomatic route with bupivacaine after bimaxillary osteotomy surgery for greater control of postoperative pain. In this way, the researchers aim to maintain the pre-incisional infiltration of LA with lidocaine plus bupivacaine and adrenaline in the surgical field performed by the surgeon with its well-known benefits and to perform the ultrasound-guided block of the maxillary nerve with bupivacaine after surgery, before extubation to prolong its effect even more in the immediate postoperative period.

The investigators use a combination of LA (lidocaine and bupivacaine) for pre-incisional infiltration of the surgical field. The combination of several local anesthetics in the same nerve block is sometimes used in perioperative anesthesia with the intention of compensating for the short duration of action of some agents with a rapid onset of action, such as lidocaine, and the high latency of agents with a longer action, such as bupivacaine. The combination of lidocaine and bupivacaine offers clinical advantages (rapid onset, long duration). This is a widespread practice among professionals in maxillofacial surgery. It is also a way to avoid the use of maximum doses of these LAs.

By performing the bilateral ultrasound-guided maxillary nerve block with bupivacaine after the surgical incision, the researchers were able to extend the effect of the nerve block for greater control of postoperative pain. Postoperative pain control is a key factor in achieving greater patient satisfaction, better rehabilitation and shorter hospital stays. Current clinical guidelines recommend the management of postoperative pain control in a multimodal manner; and this includes the use of LA for infiltration of the surgical field and the performance of peripheral nerve blocks.

To date, studies describing maxillary nerve block prior to surgeries of the middle third of the face (orthognathic surgery, cleft palate, trauma) have been described; However, there are no studies of the practice of maxillary nerve block at the end of surgery, prior to extubation. If the investigators assume that the patient receives general anesthesia (with their respective analgesics in the form of opioids, anti-inflammatories, paracetamol and other adjuvants) together with the infiltration of LA from the surgical field before starting surgery, and that this implies sufficient intraoperative analgesic coverage, the investigators propose with this study that anesthesiologists could postpone the maxillary nerve block at the end of surgery. for a greater long-term benefit of the patient in the immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled bimaxillary surgery

Exclusion Criteria:

* refusal to participate in the study
* patients scheduled for bimaxillary surgery together with another complementary surgical procedure (such as rhinoplasty, blepharoplasty)
* age < 18 years
* reinterventions
* urgent surgeries
* allergies to local anesthetics
* allergies to anti-inflammatories
* allergies to opioids
* ASA ≥3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Inmediate Postoperative pain | 2 hours postoperatively
  Postoperative pain in patients undergoing elective bimaxillary osteotomy, evaluated using the visual analog pain scale in the immediate postoperative period (2 hours postoperative). VAS: Visual analogue scale (0=minimum pain - 10=maximum pain)

SECONDARY OUTCOMES:
Pain at 8 hours postoperatively | 8 hours postoperatively
  Pain in patients undergoing elective bimaxillary osteotomy, evaluated using the visual analog pain scale at 8 hours postoperatively. VAS: Visual analogue scale (0=minimum pain - 10=maximum pain)
Pain 18 hours after surgery | 18 hours postoperatively
  Pain in patients undergoing elective bimaxillary osteotomy, evaluated using the visual analog pain scale at 18 hours postoperatively. VAS: Visual analogue scale (0=minimum pain - 10=maximum pain)
Inmediate Use of Opioids | 2 hours postoperatively
  Use of rescue opioids (milligrams of methadone) in the immediate postoperative period in resuscitation ward (milligrams of intravenous methadone at 2 hours postoperatively)
Use of rescue opioids from 2 to 18 hours postoperatively | 2 to 18 hours postoperatively
  Use of rescue oipoids in the hospitalization ward (milligrams of subcutaneous methadone from 2 to 18 hours postoperatively)
Incidence of immediate postoperative nausea and vomiting | 2 hours postoperatively
  Incidence of immediate postoperative nausea and vomiting (PONV) in resuscitation ward (2 hours postoperatively)
Incidence of postoperative nausea and vomiting up to 18 hours postoperatively | 18 hours postoperatively
  Incidence of postoperative nausea and vomiting up to 18 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Servei Central d'Anestesiologia Centro Medico Teknon, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study protocol along with the informed consents, statistical analysis and report of the ethical committee will be publicly accessible.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2024

REFERENCES:
- [Background] Brkovic B, Andric M, Calasan D, Milic M, Stepic J, Vucetic M, Brajkovic D, Todorovic L. Efficacy and safety of 1% ropivacaine for postoperative analgesia after lower third molar surgery: a prospective, randomized, double-blinded clinical study. Clin Oral Investig. 2017 Apr;21(3):779-785. doi: 10.1007/s00784-016-1831-2. Epub 2016 Apr 25. PMID 27114091
- [Background] Budharapu A, Sinha R, Uppada UK, Subramanya Kumar AV. Ropivacaine: a new local anaesthetic agent in maxillofacial surgery. Br J Oral Maxillofac Surg. 2015 May;53(5):451-4. doi: 10.1016/j.bjoms.2015.02.021. Epub 2015 Mar 24. PMID 25818492
- [Background] Cuvillon P, Nouvellon E, Ripart J, Boyer JC, Dehour L, Mahamat A, L'hermite J, Boisson C, Vialles N, Lefrant JY, de La Coussaye JE. A comparison of the pharmacodynamics and pharmacokinetics of bupivacaine, ropivacaine (with epinephrine) and their equal volume mixtures with lidocaine used for femoral and sciatic nerve blocks: a double-blind randomized study. Anesth Analg. 2009 Feb;108(2):641-9. doi: 10.1213/ane.0b013e31819237f8. PMID 19151302
- [Background] Sisk AL. Vasoconstrictors in local anesthesia for dentistry. Anesth Prog. 1992;39(6):187-93. PMID 8250339
- [Background] Mesnil M, Dadure C, Captier G, Raux O, Rochette A, Canaud N, Sauter M, Capdevila X. A new approach for peri-operative analgesia of cleft palate repair in infants: the bilateral suprazygomatic maxillary nerve block. Paediatr Anaesth. 2010 Apr;20(4):343-9. doi: 10.1111/j.1460-9592.2010.03262.x. Epub 2010 Feb 23. PMID 20199610
- [Background] Sola C, Raux O, Savath L, Macq C, Capdevila X, Dadure C. Ultrasound guidance characteristics and efficiency of suprazygomatic maxillary nerve blocks in infants: a descriptive prospective study. Paediatr Anaesth. 2012 Sep;22(9):841-6. doi: 10.1111/j.1460-9592.2012.03861.x. Epub 2012 May 15. PMID 22587691
- [Background] Chiono J, Raux O, Bringuier S, Sola C, Bigorre M, Capdevila X, Dadure C. Bilateral suprazygomatic maxillary nerve block for cleft palate repair in children: a prospective, randomized, double-blind study versus placebo. Anesthesiology. 2014 Jun;120(6):1362-9. doi: 10.1097/ALN.0000000000000171. PMID 24525630
- [Background] Bouzinac A, Tournier JJ, Dao M, Delbos A. Ultrasound-guided maxillary nerve block in adults: feasibility and efficiency for postoperative analgesia after maxillary osteotomy. Minerva Anestesiol. 2014 Jul;80(7):860-1. Epub 2014 Jan 29. No abstract available. PMID 24472751
- [Background] Wang YH, Wang DR, Liu JY, Pan J. Local anesthesia in oral and maxillofacial surgery: A review of current opinion. J Dent Sci. 2021 Oct;16(4):1055-1065. doi: 10.1016/j.jds.2020.12.003. Epub 2020 Dec 17. PMID 34484571
- [Background] Molins G, Valls-Ontanon A, De Nadal M, Hernandez-Alfaro F. Ultrasound-Guided Suprazygomatic Maxillary Nerve Block Is Effective in Reducing Postoperative Opioid Use Following Bimaxillary Osteotomy. J Oral Maxillofac Surg. 2024 Apr;82(4):412-421. doi: 10.1016/j.joms.2023.12.018. Epub 2024 Jan 2. PMID 38253318
- [Background] Gocmen G, Ozkan Y. Comparison of the Efficacy of Local Infiltration and Mandibular Block Anesthesia With Articaine for Harvesting Ramus Grafts. J Oral Maxillofac Surg. 2016 Nov;74(11):2143-2150. doi: 10.1016/j.joms.2016.05.008. Epub 2016 May 20. PMID 27294877

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT06460051/Prot_SAP_000.pdf